CLINICAL TRIAL: NCT00800358
Title: A Multi Centre, Open Label, Parallel Group, Randomized Controlled Trial to Compare the Safety and Efficacy of Oral Paricalcitol Versus Oral Calcitriol in the Treatment of Secondary Hyperparathyroidism in Dialysis Patients
Brief Title: Safety and Efficacy Study of Paricalcitol Versus Calcitriol in the Treatment of Secondary Hyperparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penang Hospital, Malaysia (Other Government)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr.Ong Loke Meng, Consultant Nephrologist, Penang Hospital, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol No: CT 08-02
Record Dates: First submitted 2008-11-30; First posted 2008-12-02 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Hyperparathyroidism; Kidney Disease
Keywords: Secondary hyperparathyroidism; End stage renal disease; Haemodialysis; Peritoneal dialysis; Paricalcitol (Zemplar); Calcitriol
MeSH Terms: conditions — Hyperparathyroidism; Kidney Diseases; Hyperparathyroidism, Secondary; Kidney Failure, Chronic | interventions — paricalcitol; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oral Paricalcitol in varying doses
  Interventions: Drug: Paricalitol
- 2 (Active Comparator): Calcitriol
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Paricalitol — oral paricalcitol variable daily dosing based on intact PTH level for 6 months
  Other Names: Zemplar
  Arms: 1
Drug: Calcitriol — oral calcitriol variable daily dosing based on intact PTH level for 6 months
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether oral paricalcitol is safer and more efficacious compared to oral calcitriol in the treatment of hyperparathyroidism in chronic kidney disease patients undergoing dialysis.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism, a common consequence of chronic kidney disease, results from abnormal regulation of calcium and phosphate homeostasis. The early administration of calcium supplements or vitamin D attenuates the development and progression of hyperparathyroidism, preventing or retarding the emergence of many of the serious complications of chronic kidney disease. However, these vitamin D derivatives also have serious side effects, including hypercalcemia and hyperphosphatemia and, as a result, a high level of the calcium-phosphate product. These adverse outcomes have prompted the development of novel, "nonhypercalcemic" vitamin D analogues. Three of these analogues have recently been marketed for clinical use in patients with chronic kidney disease: 19-nor-1,25-dihydroxyvitamin D2 (paricalcitol), 1 -hydroxyvitamin D2 (doxercalciferol), and 22-oxacalcitriol.

Oral paricalcitol was developed to provide a convenient, alternative therapy, particularly for Peritoneal Dialysis patients in whom regular intravenous administration of paricalcitol is not practical. This study is designed to determine the proportion of patients with 'End stage renal failure' on haemodialysis or peritoneal dialysis and secondary hyperparathyroidism who achieved more than 30% reduction in baseline iPTH concentration at 24 weeks of treatment with Paricalcitol or Calcitriol capsules.

ELIGIBILITY:
Inclusion Criteria:

* Age at or above 18 years
* End stage renal disease on regular maintenance haemodialysis or peritoneal dialysis for at least 3 months
* iPTH level of 300 pg/ml or greater at baseline
* Written informed consent by subject or guardian
* Female patients will either be post-menopausal for more than 2 years, surgically sterile or if of childbearing age, using double contraception

Exclusion Criteria:

* Baseline calcium value more than 2.87 mmol/L
* Baseline Ca x P of greater than 5.63 mmol2/l2
* Positive for HBsAg or Hepatitis C with raised ALT twice above upper limit of normal or evidence of liver cirrhosis
* Clinically significant gastrointestinal disease
* History of allergic reaction to calcitriol or other vitamin D compounds
* Inability or unwillingness to provide written consent.
* Inability or unwillingness to comply with the requirements of the protocol as determined by the investigator.
* Pregnancy, breastfeeding or use of non-reliable method of contraception.
* Use of medications prohibited prior to randomization such as ketoconazole and other strong P450 3A inhibitors including atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir
* Necessity for calcitonin, biphosphonates, maintenance oral or intravenous glucocorticoid or cinacalcet or other drugs that may affect calcium or bone metabolism.
* Alcohol or substance abuse within 6 months prior to screening
* Other medical condition which, in the investigator's judgement, may be associated with increased risk to the subject or may interfere with study assessments or outcomes.
* Participation in another clinical trial and/or receipt of investigational drugs within 4 weeks prior to screening visit.
* If PD subjects had active peritonitis within one month prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
More than 30% reduction in baseline iPTH concentration at 24 weeks of treatment with Paricalcitol or Calcitriol capsules. | 24 weeks

SECONDARY OUTCOMES:
Quantum of reduction in alkaline phosphatase level, Time duration to achieve the target level of iPTH. (Titration time), Serum Calcium, phosphate, Ca x Po4 product change from baseline | 24 weeks
Incidence of hypercalcaemic episodes | Through out 24 weeks of participation from the time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ong L Meng, MBBS, MRCP, Principal Investigator — Clinical Research Centre, Penang Hospital
Locations (11):
- Malaysia (11):
  - Hospital Sultanah Bahiyah Haemodialysis Unit KM 6 Jalan Langgar, Alor Star, Kedah
  - Hemodialysis Unit, Raja Perempuan Zainab II Hospital, Kota Bharu, Kelantan
  - Haemodialysis Unit, Melaka Hospital, Malacca, Melaka
  - Hemodialysis Unit, Tengku Ampuan Afzan Hospital, Kuantan, Pahang
  - Hemodialysis Unit, Taiping Hospital, Taiping, Perak
  - Clinical Research Centre, Penang Hospital, George Town, Pulau Pinang
  - Haemodialysis Unit, Seberang Jaya Hospital, Seberang Jaya, Pulau Pinang
  - Nephrology Department, Tengku Ampuan Rahimah Hospital, Klang, Selangor
  - Hemodialysis Unit, Kuala Lumpur Hospital, Kuala Lumpur, Selangor
  - Haemodialysis Unit, Serdang Hospital, Serdang, Selangor
  - Hemodialysis Unit, Tuanku Ja'afar Seremban Hospital, Seremban, Selangor

REFERENCES:
- [Derived] Ong LM, Narayanan P, Goh HK, Manocha AB, Ghazali A, Omar M, Mohamad S, Goh BL, Shah S, Seman MR, Vaithilingam I, Ghazalli R, Rahmat K, Shaariah W, Ching CH; Oral Paricalcitol in ESRD Study Group. Randomized controlled trial to compare the efficacy and safety of oral paricalcitol with oral calcitriol in dialysis patients with secondary hyperparathyroidism. Nephrology (Carlton). 2013 Mar;18(3):194-200. doi: 10.1111/nep.12029. PMID 23311404